CLINICAL TRIAL: NCT06739291
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Anti-tumor Activity and Food Effect of SIGX1094R in Patients With Advanced Solid Tumors
Brief Title: A Study of SIGX1094R in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Signet Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG-SIGX1094R-CT-001
Record Dates: First submitted 2024-12-06; First posted 2024-12-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
Keywords: Focal Adhesion Kinase inhibitor; FAK inhibitor; SIGX1094R

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SIGX1094R (Experimental): Oral SIGX1094R administered once daily.
  Interventions: Drug: SIGX1094R

INTERVENTIONS:
Drug: SIGX1094R — Single drug treatment by SIGX1094R, orally administered once daily.

SUMMARY:
This is a phase I clinical, first-in-human study of SIGX1094R monotherapy. The goal of this trial is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), anti-tumor activity and food effect of SIGX1094R in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study consists of two parts: SIGX1094R dose escalation study; food effect and SIGX1094R multiple-dose expansion study.

Part of SIGX1094R dose escalation study:

* the primary objective is to evaluate the safety and tolerability of SIGX1094R, and to define the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D).
* the secondary objective is to evaluate the PK profile and preliminary efficacy of SIGX1094R, and to explore the relationship between PD parameters and efficacy.

Part of food effect and SIGX1094R multiple-dose expansion study:

* the primary objective is to evaluate the food effect on PK profile of SIGX1094R.
* the secondary objective is to further evaluate the anti-tumor activity, safety and tolerability of SIGX1094R, and to further evaluate the relationship between PD parameters and efficacy.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria before being enrolled in the study.

1. Patients must be able to understand the procedures and methods of this clinical study, voluntarily participate in the study and sign the ICF.
2. Patients aged ≥18 years when signing the ICF, male or female.
3. Patients with histologically, cytologically, or clinically proven advanced solid tumors (locally advanced or metastatic) that do not have standard treatment available, have disease progression on/after standard treatment, or cannot tolerate standard treatment.
4. Patients with at least one evaluable tumor lesion according to the RECIST v1.1; patients who have no measurable lesions but have evaluable lesions are allowed to be enrolled as judged by the investigator.
5. Patients (according to patients' option) will provide a pre-treatment tumor specimen (archival or fresh biopsy samples). If a fresh biopsy is required, procedures more invasive than a core biopsy or significant risk procedures for which the procedure-associated absolute risk of mortality or major morbidity in the patient's clinical setting and specific institution is 2% or higher, should not be utilized. The tumor tissue is used for pFAK status confirmation, without restriction on enrollment.
6. ECOG score ≤ 1.
7. Life expectancy ≥ 3 months
8. Patients with adequate organ function, including:

   * Liver function (no history of liver protection therapy 7 days before screening): total bilirubin (TBIL) ≤ 1.5×ULN, alanine aminotransferase (ALT)

     * 3×ULN, aspartate aminotransferase (AST) ≤ 3×ULN (no liver metastasis); if there is liver metastasis, ALT and AST ≤ 5×ULN; albumin ≥ 30 g/L.
   * Renal function: Creatinine clearance ≥ 50 mL/min (calculated according to Cockcroft-Gault formula).
   * Hematology (no blood transfusion or hematopoietic stimulating factor treatment within 14 days; no treatment with erythropoietin or thrombopoietin within 7 days): absolute neutrophil count (ANC) ≥ 1.5×10^9/L, platelet (PLT) ≥ 100×10^9/L, and hemoglobin (Hb) ≥ 90 g/L.
   * Coagulation function: activated partial thromboplastin time ≤ 1.5 × ULN and international normalized ratio ≤ 1.5 × ULN.
9. Women of reproductive age must have a negative blood pregnancy test result within 7 days prior to the first dose and promise to adhere to fully effective contraception or abstinence from the beginning of the screening period until 6 months after the last dose of study treatment; male patients must promise to adhere to fully effective contraception or abstinence from the beginning of the screening period until 6 months after the last dose of study treatment.

Exclusion Criteria:

Patients who meet any of the following criteria cannot be enrolled in this study.

1. Patients with hypersensitivity to the active ingredient or excipient ingredient of SIGX1094R, or a history of severe allergy.
2. Patients who have received cytotoxic chemotherapeutic drugs or small molecule targeted drugs within 4 weeks prior to the first dose. Note: For mitomycin C or nitrosoureas, 6-week washout is required; for small-molecule targeted drugs and oral fluorouracil drugs, a washout period of 2 weeks or 5 T1/2 of the drug (whichever is shorter) is required.
3. Anti-tumor endocrine therapy, radiotherapy, interventional embolization, radiofrequency, proton therapy, radioimmunotherapy, immunotherapy or other biotherapies within 4 weeks prior to the first dose (if 5 T1/2 of the drug/therapy used by the patient is confirmed to be < 4 weeks, 5 T1/2 shall prevail).
4. Patients who have received anti-tumor treatment with medicine/proprietary medicine within 2 weeks prior to the first dose. Note: This criterion is relevant to China study only.
5. Patients who have received other clinical investigational drugs or therapies that are not on the market within 4 weeks or 5 T1/2 prior to the first dose, whichever is longer.
6. Prior treatment with focal adhesion kinase (FAK) inhibitors.
7. Patients who have received moderate-to-strong cytochrome P450(CYP)3A4, CYP3A5 inhibitors, or moderate-to-strong CYP3A4 or CYP3A5 inducers, or moderate-to-strong P-gp and BCRP inhibitors, within 14 days prior to the first dose. Note: please see the https://www.fda.gov/drugs/drug- interactions labeling/drug-development-and-drug-interactions-table- substrates inhibitors-and-inducers for the Inhibitors and Inducers of the CYP enzyme or transporters.
8. Patients who have received an anti-acid drug or gastric acid reducing agents within 14 days prior to the first dose and cannot be discontinued for the duration of the study.
9. Pregnant or lactating women.
10. Patients whose adverse reactions of prior anti-tumor therapy assessed according to CTCAE v5.0 at the time of screening have not returned to Grade ≤ 1 (except for toxicities that are of no safety risk as judged by the investigator, such as alopecia, gasping, γ-glutamyl transferase (GGT) increased, Alkaline phosphatase (ALP) increased, grade 2 peripheral neurotoxicity, and decreased thyroid function stabilized by hormone replacement therapy).
11. Presence of clinically symptomatic metastases to central nervous system or meninges or other evidence showing that metastatic lesions in central nervous system or meninges have not yet been controlled at screening, which, at the investigator's discretion, is not suitable for enrollment. Note: Patients with central nervous system or meningeal metastases who are asymptomatic or stable after treatment prior to the first dose may be considered for enrollment.
12. A history of severe neurological or psychiatric disorders, including epilepsy, dementia, and moderate to severe depression.
13. History of drug abuse or dependence.
14. Clinically serious and uncontrolled cardiovascular diseases, including:

    * Serious arrhythmia or conduction abnormality at screening, such as ventricular arrhythmia that requires clinical intervention, atrioventricular block II-III degree, etc.
    * Myocardial infarction within 12 months prior to the first dose.
    * Acute coronary syndrome, placement of stents for stable or unstable angina pectoris, cardiac failure congestive, aortic dissection, cerebral stroke or other Grade ≥ 3 cardiovascular and cerebrovascular events within 6 months prior to the first dose.
    * Patients who have had arterial or deep vein thrombosis within 6 months prior to the first dose, or patients requiring international normalized ratio (INR) monitoring or using anticoagulants at the time of screening; patients with hemorrhagic diseases, active ulcer, and experienced gastrointestinal perforation. Note: Patients with superficial venous thrombosis who do not require treatment may be considered for enrollment; patients who are able to stop anticoagulants within 2 weeks prior to the first dose and during medication may be considered for enrollment.
    * Patients with average QTcF of triplicate 12-lead ECGs at screening > 470ms [Note: QTcF is calculated according to Fridericia formula, QTcF= QT/(RR^0.33)].
    * Patients with any risk factors that may prolong the QTc interval, such as uncorrectable hypokalemia, hereditary long QT syndrome, and the use of medications that prolong the QTc interval (primarily Class Ia, Ic, and III antiarrhythmic drugs).
    * Patients with New York Heart Association (NYHA) Class ≥ II cardiac failure at screening.
    * Left ventricular ejection fraction (LVEF) < 50% at screening.
    * Hypertension (defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) which has not been consistently controlled with medication at screening.
15. Patients with hyperglycemia that cannot be stably controlled with medication at screening.
16. Patients with pulmonary embolism within 6 months prior to the first dose, or interstitial pneumonia at screening.
17. Prior allogeneic stem cell transplantation, bone marrow transplantation or vital organ transplantation.
18. Patients who have undergone surgery on vital organs (other than aspiration biopsy) or suffered major trauma within 4 weeks prior to the first dose, or patients who have not recovered from any surgical effect at screening, or who are scheduled for major surgery during the study period.
19. Patients with uncontrolled infectious diseases, congenital immunodeficiency diseases, acquired immunodeficiency syndrome [human immunodeficiency virus antibody (HIV-Ab) positive], syphilis (syphilis antibody-positive), or active hepatitis B [hepatitis B virus (HBV) - deoxyribonucleic acid (DNA) >500 IU/ml]; hepatitis C virus (HCV) infection (HCV antibody positive and HCV ribonucleic acid amplification quantitative test positive). Patients with well controlled HIV, HBV, and HCV infections may be enrolled with no significant safety risk in the judgment of the investigator; see https://www.fda.gov/media/121319/download for definition of well controlled.
20. Patients with severe active infection, including but not limited to bacteremia and severe pneumonia within 2 weeks prior to the first dose; patients with an active infection requiring intravenous antibiotics within 2 weeks prior to the first dose.
21. Patients with conditions that may affect drug absorption as judged by the investigator, such as dysphagia, chronic diarrhea, or prior small bowel resection.
22. Patients with active autoimmune diseases, such as rheumatic disorder and rheumatoid disease.
23. The investigator considers that the patient is not suitable for participating in this study (e.g., study drug is not in the best interest of patient, patients with mental disorder, patients with poor compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From the first dose to 28 days after the last dose. Last for approximately 18 months.
  To evaluate the safety and tolerability of SIGX1094R. AEs will be evaluated per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE),Version 5.0.
Incidence of serious adverse events (SAEs) | From the first dose to 28 days after the last dose. Last for approximately 18 months.
  To evaluate the safety and tolerability of SIGX1094R. SAEs will be evaluated per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE),Version 5.0.
Abnormalities or changes in laboratory tests | Approximately 18 months
  To evaluate the safety and tolerability of SIGX1094R.
Abnormalities or changes in vital signs | Approximately 18 months
  To evaluate the safety and tolerability of SIGX1094R.
Abnormalities or changes in electrocardiograms (ECGs) | Approximately 18 months
  To evaluate the safety and tolerability of SIGX1094R.
Abnormalities or changes in physical examinations | Approximately 18 months
  To evaluate the safety and tolerability of SIGX1094R.
Abnormalities or changes in Eastern Oncology Collaborative Group (ECOG) scores | Approximately 18 months
  To evaluate the safety and tolerability of SIGX1094R.
Incidence of dose-limiting toxicity (DLT) events | From the first treatment of single dosing (5 days in single dosing period ) to the end of Cycle 1 (21 days a Cycle in multiple dosing period ).
  Collect the incidence, classification, severity, and frequency of DLT. To evaluate the safety and tolerability of SIGX1094R.
Maximum tolerated dose (MTD) | Approximately 18 months
  To determine the MTD of SIGX1094R.
Recommended phase 2 dose (RP2D) | Approximately 18 months
  To determine the RP2D of SIGX1094R.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Time points at Day 1 to Day 5 in single-dose period. Time points at Cycle 1 Day1, Cycle 1 Day 8, Cycle 1 Day15, Cycle 1 Day 21 in Cycle 1, and Cycle n Day 1 from Cycle 2, in multiple-dose period. Each Cycle is 21 days.
  To assess pharmacokinetics (PK) of SIGX1094R in plasma following a single and multiple doses of SIGX1094R.
Time of maximum observed concentration (Tmax) | Time points at Day 1 to Day 5 in single-dose period. Time points at Cycle 1 Day1, Cycle 1 Day 8, Cycle 1 Day15, Cycle 1 Day 21 in Cycle 1, and Cycle n Day 1 from Cycle 2, in multiple-dose period. Each Cycle is 21 days.
  To assess PK of SIGX1094R in plasma following a single and multiple doses of SIGX1094R.
Area under the concentration-time curve (AUC) | Time points at Day 1 to Day 5 in single-dose period. Time points at Cycle 1 Day1, Cycle 1 Day 8, Cycle 1 Day15, Cycle 1 Day 21 in Cycle 1, and Cycle n Day 1 from Cycle 2, in multiple-dose period. Each Cycle is 21 days.
  To assess PK of SIGX1094R in plasma following a single and multiple doses of SIGX1094R.
Half-life (t1/2) | Time points at Day 1 to Day 5 in single-dose period. Time points at Cycle 1 Day1, Cycle 1 Day 8, Cycle 1 Day15, Cycle 1 Day 21 in Cycle 1, and Cycle n Day 1 from Cycle 2, in multiple-dose period. Each Cycle is 21 days.
  To assess PK of SIGX1094R in plasma following a single and multiple doses of SIGX1094R.
Objective response rate (ORR) | Approximately 18 months
  Proportion of subjects whose best response is observed to be complete response (CR) or partial response (PR) throughout the study. Assessed by RECIST 1.1 criteria.
Progression-free survival (PFS) | Approximately 18 months
  Time from Day 1 of treatment with the study drug to progressive disease (PD) or death from any cause. Assessed by RECIST 1.1 criteria.
Duration of response (DOR) | Approximately 18 months
  Time from first tumor assessment of CR or PR on study treatment to first assessment of PD or death due to any cause. Assessed by RECIST 1.1 criteria.
Overall survival (OS) | Approximately 18 months
  Time from Day 1 of treatment with the study drug to death from any cause. Assessed by RECIST 1.1 criteria.
Disease control rate (DCR) | Approximately 18 months
  Proportion of subjects whose best response is observed to be CR, PR, or stable disease (SD) (duration ≥ 12 weeks) throughout the study. Assessed by RECIST 1.1 criteria.
Clinical benefit rate (CBR) | Approximately 18 months
  Proportion of subjects whose best response is observed to be CR, PR, or SD (duration ≥ 24 weeks) throughout the study.
Changes of phosphorylated Focal Adhesion Kinase (pFAK) in tumor tissues | Baseline to approximately 18 months
  Determine the changes of phosphorylated Focal Adhesion Kinase (pFAK) from baseline in tumor tissues and assess its relationship with efficacy.

OTHER OUTCOMES:
22. Changes of circulating tumor DNA (ctDNA) | Baseline to approximately 18 months
  Determine the changes of ctDNA from baseline in blood and assess its relationship with efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided